CLINICAL TRIAL: NCT05651893
Title: Efficacy of Second Forward-view Examination of Left Colon for Adenoma Detection During Colonoscopy: a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Efficacy of Second Forward-view Examination of Left Colon for Adenoma Detection During Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: No.85 Hospital, Changning, Shanghai, China (Other); Shanxi Provincial People's Hospital (Other Government); The General Hospital of Eastern Theater Command (Other); The Sixth Affiliated Hospital of Guangzhou Medical University (Other); Fudan University (Other); Kunshan Hospital of Traditional Chinese Medicine (Unknown); Ningjin County Hospital (Unknown); Qinghai People's Hospital (Other); The First Affiliated Hospital of Yangtze University (Other); Qujing NO.1 Hospital (Unknown); Jiangxi Provincial People's Hopital (Other); Yueyang Central Hospital (Other); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); The First People's Hospital of Changde City (Other); Xuzhou Central Hospital (Other); Wenzhou Central Hospital (Other); Anhui Provincial Hospital (Other Government); Jiangsu Provincial People's Hospital (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, MD,Director, Head of Department of Gastroenterology and Digestive Endoscopy Center, Principal Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SFW2022-01
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Colon Adenoma
Keywords: Adenoma detection rate; colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second forward view examination group (Experimental): After successful intubation of the cecum, the colonoscope is withdrawn to the splenic curvature with the colonic mucosa carefully inspected. Then the left colon, including the splenic curvature to the anus, is examined twice in the forward view.
  Interventions: Behavioral: re-examination
- Extended withdrawal time group (Experimental): After successful intubation of the cecum, the colonoscope is withdrawn to the splenic curvature with the colonic mucosa carefully inspected. The colonoscope was withdrawn to the anus directly with withdrawal time extended to the double routine withdrawal time of the left colon.
  Interventions: Behavioral: extended withdraw time

INTERVENTIONS:
Behavioral: re-examination — During colonoscopy, the left colon was examined a second time in the forward view.
  Arms: Second forward view examination group
Behavioral: extended withdraw time — During colonoscopy, the left colon was examined with double basic withdrawal time in the forward view.
  Arms: Extended withdrawal time group

SUMMARY:
The incidence of colorectal cancer in China is increasing year by year. Studies have shown that colorectal cancer is more common in the left colon，especially in the China. Our previous study also showed a higher rate of missed adenoma in the left colon than the right colon during colonoscopy. Additionally, prolonging withdrawal time could only improve the ADR of right colon, but had limited effect on the ADR of left colon in our previous research. Our aim is to evaluate the effect of a second forward view examination of the left colon on the detection of adenoma detection during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age are between 40-75, or aged 76-85 depending on his condition
* Patients who have indications for screening
* Patients who have signed inform consent form.

Exclusion Criteria:

* Patients who have undergone colonic resection
* Patients with alarming signs and symptoms of colorectal cancer: hematochezia, melena, anemia, weight loss, abdominal mass, positive digital rectal examination
* Patients with abnormal blood coagulation or taking antiplatelets or anticoagulants within 7 days before colonoscopy
* Patients with inflammatory bowel diseases
* Patients with a history of abdominal surgery, or highly suspected or confirmed colorectal cancers by radiographic and laboratory tests Patients with hereditary colorectal cancer syndrome (including familial adenomatous polyposis).
* Patients with pregnancy, severe chronic cardiopulmonary and renal disease.
* Patients with failed cecal intubation
* Patients with poor BPQ that necessitated a second bowel preparation
* Patients with therapeutic colonoscopy for existing lesions
* Patients refusing to participate or to provide informed consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1516 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Left colon adenoma detection rate (LCADR) | 60 minutes
  LCADR is the number of patients with at least one adenoma in the left colon, divided by the total number of patients.

SECONDARY OUTCOMES:
adenoma detection rate(ADR) | 60 minutes
  ADR is the number of patients with at least one adenoma, divided by the total number of patients.
left colon adenomas per colonoscopy (LCAPC) | 60 minutes
  LCAPC was calculated as the number of adenomas detected during in left colon colonoscopy withdraw divided by the number of colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Background] Zhao S, Yang X, Wang S, Meng Q, Wang R, Bo L, Chang X, Pan P, Xia T, Yang F, Yao J, Zheng J, Sheng J, Zhao X, Tang S, Wang Y, Wang Y, Gong A, Chen W, Shen J, Zhu X, Wang S, Yan C, Yang Y, Zhu Y, Ma RJ, Wang R, Ma Y, Li Z, Bai Y. Impact of 9-Minute Withdrawal Time on the Adenoma Detection Rate: A Multicenter Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e168-e181. doi: 10.1016/j.cgh.2020.11.019. Epub 2020 Nov 19. PMID 33220526
- [Background] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046